CLINICAL TRIAL: NCT05238623
Title: Imbalances of Regional Pulmonary Ventilation in Patients With Post-acute-COVID-19 Symptoms
Brief Title: Imbalances of Regional Pulmonary Ventilation in Patients With Post-acute-COVID-19
Status: Not yet recruiting | Type: Observational
Sponsor: Jan-Christoph Lewejohann (Other)
Responsible Party: Sponsor-Investigator, Jan-Christoph Lewejohann, Investigator, Jena University Hospital
Organization: Jena University Hospital (Other)
Other Study IDs: KIM-IV-EIT03
Record Dates: First submitted 2022-02-08; First posted 2022-02-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: COVID-19 Pneumonia; Post-acute COVID-19 Syndrome; Electric Impedance
Keywords: Electric Impedance; CT; Tomography; regional ventilation; post-acute-COVID-19 syndrome; post-COVID-19; EIT; electroimpedance tomography; long-COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control cohort: lung-healthy volunteers get a EIT measurement
- Case cohort: Patients who receive standard CT and pulmonary function testing also receive electroimpedance tomography measurement
  Interventions: Diagnostic Test: additional EIT Measurement

INTERVENTIONS:
Diagnostic Test: additional EIT Measurement — Patients who receive standard CT and pulmonary function testing also receive electroimpedance tomography measurement. The lunghealthy Patients in the control group only receive a EIT.
  Groups: Case cohort

SUMMARY:
Investigation of the correlation of CT-morphological changes of the lung compared to regional ventilation distribution on electrical impedance tomography in patients with post-acute-Covid-19 symptoms.

DETAILED DESCRIPTION:
Prospective non-interventional, monocentric observational study on imbalances in regional lung ventilation compared to chest CT in post-acute-Covid-19. The aim is to verify the agreement between computerized tomography derived imaging variables and electrical impedance tomography in detecting lung ventilation imbalances. The primary study objective is to match CT morphological changes in regional ventilation in post-acute-COVID-19 patients and/or changes in lung function examination, with changes that can be visualized by electroimpedance tomography.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing a Chest CT due to suspected post-acute-Covid-19-syndrome
* >18 years
* informed consent.

Exclusion Criteria:

* trauma patients and patients with unstable spinal injuries or fractures
* patients with an BMI over 50
* patients with uncontrolled body movements
* Patients with a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the post-COVID-19 outpatient clinic are screened.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between tomography and electroimpedance tomography | until May 2022
  The primary study objective is to match CT morphological changes in regional ventilation in post-COVID patients and/or changes in lung function examination with changes that can be visualized by electroimpedance tomography.

SECONDARY OUTCOMES:
Correlation between lung function testing and electroimpedance tomography | until May 2022

CONTACTS AND LOCATIONS:
Overall Officials: Phillip A Reuken, Dr., Study Director — Jena University Hospital, Klinik für Innere Medizin IV
Locations (1):
- Klinik für Notfallmedizin, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT05238623/Prot_SAP_000.pdf